CLINICAL TRIAL: NCT00467194
Title: A Phase I Study of Rapamycin in Combination With Bevacizumab in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Sirolimus and Bevacizumab in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Choo Su Pin, Senior Consultant, National Cancer Centre, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540163; SINGAPORE-06-17-HEP
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; advanced adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sirolimus; Bevacizumab

ARMS (1):
- Phase I study of rapamycin and bevacizumab (Experimental): Rapamycin (available as 1mg per tablet; Wyeth) will be given orally once in the morning before meal. The starting dose of rapamycin will be 1mg administered once daily. All doses of rapamycin will be preceded by an oral loading dose three times the maintenance dose on day 1. The dose of rapamycin will be increased at each dose level.
  Bevacizumab (100mg/4ml; Roche) will start concurrently with rapamycin. It will be diluted in a total of 100ml of 0.9% sodium chloride given via intravenous injection. The first dose will be infused over 90 minutes. If the first infusion is tolerated without any adverse infusion-related events (fever and/or chills), the second infusion may be delivered over 60 minutes. If the 60- minute infusion is well tolerated, the subsequent doses may be delivered over 30 minutes.
  Interventions: Drug: Rapamycin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Rapamycin
Drug: Bevacizumab

SUMMARY:
RATIONALE: Sirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab and sirolimus may also stop the growth of liver cancer by blocking blood flow to the tumor. Giving sirolimus together with bevacizumab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of sirolimus when given together with bevacizumab in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of sirolimus used in combination with bevacizumab in patients with unresectable hepatocellular carcinoma.
* Determine the toxicity profile of this regimen in these patients.

Secondary

* Determine the clinical activity of this regimen in these patients.
* Determine the pharmacokinetics of sirolimus in these patients.
* Determine the biologically active dose range of sirolimus in these patients.
* Correlate phosphorylated p70S6K activity with clinical response in patients treated with this regimen.
* Correlate PTEN, 4EBP-1, phosphorylated p70S6K, CD31, and vascular endothelial growth factor expression with clinical response in patients treated with this regimen.
* Correlate the degree of angiogenesis (as measured by DCE-CT scan) with drug levels and clinical response.

OUTLINE: This is a dose-escalation study of sirolimus.

Patients receive bevacizumab IV over 30-90 minutes once every 2 weeks and oral sirolimus once daily. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of sirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Six additional patients receive treatment at the MTD.

Blood samples are collected from healthy participants to measure p70S6 kinase activity. Patients undergo blood sample collection at baseline and periodically during study for pharmacokinetic and p70S6K activity assessment. Samples are also analyzed by high-performance liquid chromatography and tandem mass spectrophotometry to determine peak drug concentrations. Patients without archived tumor samples undergo tumor tissue biopsy at baseline. Samples are analyzed for PTEN, 4E-BP1, vascular endothelial growth factor, epidermal growth factor, p70S6K, and CD31 by immunohistochemistry. Patients also undergo DCE-CT scan at baseline and on day 29 to assess angiogenesis.

After completion of study treatment, patients are followed for 52 weeks.

PROJECTED ACCRUAL: A total of 36 patients and 5 healthy participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Histologically confirmed unresectable hepatocellular carcinoma, meeting all of the following criteria:

    * Failed 0-2 lines of chemotherapy
    * Child-Pugh class A or B for liver cirrhosis
    * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm with conventional techniques or ≥ 10 mm with spiral CT scan
    * No known brain metastases
    * Bone metastases allowed provided other measurable disease is present
  * Healthy participant

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 or Karnofsky PS 70-100%
* Life expectancy > 3 months
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* AST and ALT ≤ 5 times ULN
* Creatinine normal
* PTT < 1.5 times ULN
* Fasting serum cholesterol ≤ 350 mg/dL
* Triglycerides ≤ 300 mg/dL
* Proteinuria < 2+ by urine dipstick OR urine protein ≤ 1 g by 24-hour urine collection
* No history of allergic reactions to compounds of similar chemical or biologic composition to sirolimus or bevacizumab
* No prior thromboembolic disease that may result in bleeding or clotting problems related to use of bevacizumab including, but not limited to, the following:

  * Esophageal varices
  * Bleeding disorders
  * Deep vein thromboses
* No history of hematemesis or hemoptysis
* No other uncontrolled illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude study participation
* No HIV positivity
* Able to take oral medications
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during the course of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 28 days since prior surgery and recovered
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent traditional Chinese medicine(s)
* No concurrent long term anticoagulation with heparin or warfarin
* Concurrent prophylactic low-dose acetylsalicylic acid for patients at risk of an arterial thromboembolic event allowed
* Hepatitis B carriers must be on lamivudine during and for 6 months after completion of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-12; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 3 years
Maximum tolerated dose | 3 years

SECONDARY OUTCOMES:
Response rate (complete and partial response and stable disease) | 3 years
Progression-free survival | 3 years
Overall survival | 3 years
Distribution of p70S6K activity in peripheral blood mononuclear cells | 3 years
Correlation of p70S6K with tumor response | 3 years
Expression of tumor tissue biomarkers (PTEN, 4EBP-1, CD31, p70S6K, and vascular endothelial growth factor) | 3 years
Correlation of tumor biomarkers with response | 3 years
Best overall response (complete and partial response; stable and progressive disease) | 3 years
Change in DCE-CT scan assessment of angiogenesis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Choo Su Pin, MD, Principal Investigator — National Cancer Centre, Singapore; Toh Han Chong, MD, MBBS, MRCP, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre - Singapore, Singapore
  - Johns Hopkins Singapore International Medical Centre, Singapore

REFERENCES:
- [Background] Treiber G. mTOR inhibitors for hepatocellular cancer: a forward-moving target. Expert Rev Anticancer Ther. 2009 Feb;9(2):247-61. doi: 10.1586/14737140.9.2.247. PMID 19192962
- [Derived] Choo SP, Chowbay B, Ng QS, Thng CH, Lim C, Hartono S, Koh TS, Huynh H, Poon D, Ang MK, Chang S, Toh HC. A Phase 1 dose-finding and pharmacodynamic study of rapamycin in combination with bevacizumab in patients with unresectable hepatocellular carcinoma. Eur J Cancer. 2013 Mar;49(5):999-1008. doi: 10.1016/j.ejca.2012.11.008. Epub 2012 Dec 19. PMID 23265712